CLINICAL TRIAL: NCT02469714
Title: Integrated Care & Patient Navigators for Latinos With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Institute of Technology (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Trilogy Inc. Behavioral Healthcare (Other)
Responsible Party: Principal Investigator, Patrick Corrigan, Distinguished Professor of Psychology, Illinois Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PCORI-AD1306-01419
Record Dates: First submitted 2015-06-05; First posted 2015-06-11 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Mental Disorders
Keywords: Patient Navigator; Integrated Care; Latino; Mental health and wellness; Physical health and wellness
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Navigator Intervention (Experimental): Integrated care with a peer navigator to be provided for one year, where data will be collected at baseline, 4, 8 and 12 months.
  Interventions: Behavioral: Peer Navigator Intervention
- Controlled (No Intervention): Integrated care without a peer navigator, where data will be collected at baseline, 4, 8 and 12 months

INTERVENTIONS:
Behavioral: Peer Navigator Intervention — Peer navigators will be Hispanics/Latinos with a mental illness in recovery who will complete and meet certification for the peer navigator training program that will be evolved out of the mixed methods process. Investigators propose the peer navigators will enhance patient engagement in integrated care which will, in turn, improve physical and mental health and wellness of patients in this group
  Other Names: Peer Navigator
  Arms: Peer Navigator Intervention

SUMMARY:
The health care needs of people with serious mental illness are exacerbated by ethnic health disparities. Latinos with serious mental illness show significant health problems compared to other ethnic groups. Therefore, this project is to develop a meaningful peer-navigator program for Latinos with serious mental illness using community-based participatory research (CBPR). Investigators are currently working with seven Hispanic/Latinos with a mental illness that have formed a Consumer Research Team (CRT) that will guide this project. This project will identify and define the problem by conducting a mixed methods research thru qualitative interviews with various stakeholders defined by the investigator's CRT group. The qualitative findings will then be cross-validated in a quantitative survey by 100 Hispanic/Latinos with mental illness. This information will then be used to design an intervention using an integrated care model for Peer-Navigators. Feasibility, accessibility , acceptability and impact of the peer-navigator program will be then evaluated in a randomized control trial (RCT) with 100 Latinos with serious mental illness who will complete measures of physical health, mental health, service use and engagement at baseline, 4, 8, and 12 months. Investigators expect to show physical health improvement with the greater engagement observed in the peer navigator group. Investigators expect a similar improvement in mental health and quality of life as physical health concerns are diminished.

DETAILED DESCRIPTION:
Latinos with serious mental illnesses have an inordinately high rate of physical illness leading to a significantly shortened life. One reason is the difficulty in engaging this disenfranchised group in primary care. Integrated services through community-based outreach and care coordination are an innovative and evidence-based practice that improves physical health. Unfortunately, social determinants of health for Latinos are often a barrier to participation in integrated care. Peer navigators offer a strategy that might help members of this group. Peer navigators, in this study, are Latinos with past history of serious mental illness specially trained to help patients meet their health needs. The program will be developed through community-based participatory research (CBPR) representing a hands-on partnership between investigators and a community advisory board made up of patient partners. Given this, investigators aim to do the following. (1) Develop a peer navigator program meant to enhance the impact of already existing integrated services for Latinos with serious mental illness. (2) Using an experimental design, test the impact of peer navigators, compared to existing integrated services alone, on engagement of Latinos with serious mental illness in primary care services. This includes indices of care seeking, appointments, and satisfaction with engagement. Investigators expect these indices to be higher in the group with peer navigators. (3) Determine the comparative impact of peer navigators versus integrated-care-as-usual on subsequent health. Investigators expect to show physical health improvement with the greater engagement observed in the peer navigator group. Investigators expect a similar improvement in mental health and quality of life as physical health concerns are diminished. This proposal represents the partnership between researchers from the Center on Adherence and Self-Determination (a National Institute of Mental Health-funded Center dedicated to understanding service engagement among people with serious mental illness and their health care system) and Trilogy. Consistent with other projects, investigators will develop a Community Advisory Board to conduct CBPR and complete a mixed-methods research project to inform the peer navigator program. Based on a power-analysis, investigators will recruit 100 Latinos with serious mental illness who will complete baseline measures of physical health, mental health, service use and engagement in the previous year, quality of life, and current housing/employment status. Patients will then be randomized to an existing integrated care program for Hispanic/Latinos with mental illness with or without peer navigators for one year. Measures will be repeated at 4, 8, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Identify ethnicity as Hispanic/Latino
* Identify with experience with a mental illness

Exclusion Criteria:

* Must be 18 years or older
* Have case manager they met on a regular basis (every week for the past 4 months) for physical health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Corrigan, Psy.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

REFERENCES:
- [Background] Corrigan PW. Consumer satisfaction with institutional and community care. Community Ment Health J. 1990 Apr;26(2):151-65. doi: 10.1007/BF00752392. PMID 2191833
- [Background] Corrigan PW, Jakus MR. The Patient Satisfaction Interview for partial hospitalization programs. Psychol Rep. 1993 Apr;72(2):387-90. doi: 10.2466/pr0.1993.72.2.387. PMID 8488222
- [Background] Fischer EH, Turner JL. Orientations to seeking professional help: development and research utility of an attitude scale. J Consult Clin Psychol. 1970 Aug;35(1):79-90. doi: 10.1037/h0029636. No abstract available. PMID 5487612
- [Background] Johansen R, Hestad K, Iversen VC, Agartz I, Sundet K, Andreassen OA, Melle I. Cognitive and clinical factors are associated with service engagement in early-phase schizophrenia spectrum disorders. J Nerv Ment Dis. 2011 Mar;199(3):176-82. doi: 10.1097/NMD.0b013e31820bc2f9. PMID 21346488
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837
- [Background] Rogers ES, Ralph RO, Salzer MS. Validating the empowerment scale with a multisite sample of consumers of mental health services. Psychiatr Serv. 2010 Sep;61(9):933-6. doi: 10.1176/ps.2010.61.9.933. PMID 20810594
- [Background] Corrigan PW, Faber D, Rashid F, Leary M. The construct validity of empowerment among consumers of mental health services. Schizophr Res. 1999 Jul 27;38(1):77-84. doi: 10.1016/s0920-9964(98)00180-7. PMID 10427613
- [Background] Corrigan PW, Giffort D, Rashid F, Leary M, Okeke I. Recovery as a psychological construct. Community Ment Health J. 1999 Jun;35(3):231-9. doi: 10.1023/a:1018741302682. PMID 10401893
- [Background] Corrigan PW, Salzer M, Ralph RO, Sangster Y, Keck L. Examining the factor structure of the recovery assessment scale. Schizophr Bull. 2004;30(4):1035-41. doi: 10.1093/oxfordjournals.schbul.a007118. PMID 15957202
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] de Vet HC, Ader HJ, Terwee CB, Pouwer F. Are factor analytical techniques used appropriately in the validation of health status questionnaires? A systematic review on the quality of factor analysis of the SF-36. Qual Life Res. 2005 Jun;14(5):1203-18; dicussion 1219-21, 1223-4. doi: 10.1007/s11136-004-5742-3. PMID 16047498
- [Background] Lehman AF. The well-being of chronic mental patients. Arch Gen Psychiatry. 1983 Apr;40(4):369-73. doi: 10.1001/archpsyc.1983.01790040023003. PMID 6838316
- [Background] Lehman AF. The effects of psychiatric symptoms on quality of life assessments among the chronic mentally ill. Eval Program Plann. 1983;6(2):143-51. doi: 10.1016/0149-7189(83)90028-9. PMID 10265063
- [Background] Corrigan PW, Buican B, McCraken S. The needs and resources assessment interview for severely mentally ill adults. Psychiatr Serv. 1995 May;46(5):504-5. doi: 10.1176/ps.46.5.504. PMID 7627679
- [Background] Contopoulos-Ioannidis DG, Karvouni A, Kouri I, Ioannidis JP. Reporting and interpretation of SF-36 outcomes in randomised trials: systematic review. BMJ. 2009 Jan 12;338:a3006. doi: 10.1136/bmj.a3006. PMID 19139138
- [Background] Corrigan PW, Jakus MR. The reliability of severely mentally ill patients' report of treatment satisfaction. International Journal of Methods in Psychiatric Research 3: 215-219, 1993.
- [Background] Corrigan PW, Michaels PJ. Perceived availability of services scale. Chicago: CASD. 2012.
- [Background] Lehman AF. A quality of life interview for the chronically mentally ill. Evaluation and Program Planning 11(1): 51-62, 1988.
- See also: Projects led by Dr. Patrick Corrigan that address health disparities — http://www.chicagohealthdisparities.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 8/24/2015 to 11/20/2015. Locations for recruitment included: Trilogy, National Alliance on Mental Illness Chicago, social service providers, community coalitions, religious organizations, health fairs, and health centers that provided free or sliding scale access to care.
Pre-assignment Details: No enrolled participants (from Baseline) were excluded from the study before or after assignment to groups
Period: Overall Study
Arm/Group | Peer Navigator Intervention | Controlled
Started (Baseline) | 55 | 55
4 Month Follow-Up | 50 | 51
8 Month Follow-Up | 49 | 50
Completed (12 Month Follow-Up) | 47 | 50
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Navigator Intervention | Controlled | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.56 (9.927) | 42.67 (11.918) | 45.62 (11.311)
Sex/Gender, Customized [Number; unit: participants]
  Female | 28 | 36 | 64
  Male | 26 | 18 | 44
  Transgender | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants were required to be of Hispanic/Latino origin
  Participants
    Hispanic or Latino | 55 | 55 | 110
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 16 | 33
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 34 | 35 | 69
Language [Number; unit: participants]
  Preferred English | 16 | 25 | 41
  Preferred Spanish | 39 | 30 | 69
Education [Number; unit: participants]
  Less than High School or GED | 23 | 16 | 39
  High School or GED | 13 | 15 | 28
  Some College | 9 | 15 | 24
  Associate's Degree | 3 | 3 | 6
  Bachelor's Degree | 5 | 3 | 8
  More than a Bachelor's Degree | 2 | 3 | 5
Employment [Number; unit: participants]
  Yes | 16 | 19 | 35
  No | 39 | 36 | 75
Diagnosis [Number; unit: participants]
  Major Depression | 32 | 40 | 72
  Bipolar Disorder | 2 | 6 | 8
  Anxiety Disorder | 17 | 6 | 23
  Post Traumatic Stress | 1 | 1 | 2
  Schizophrenia | 3 | 0 | 3
  Schizoaffective | 0 | 1 | 1
  Adult ADD | 0 | 1 | 1
Sexual Orientation [Number; unit: participants]
  Heterosexual | 46 | 46 | 92
  Homosexual | 2 | 2 | 4
  Bisexual | 4 | 3 | 7
  Queer | 2 | 3 | 5
  Other | 1 | 0 | 1
  Refuse to answer | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Weekly Health Appointment Measure
Description: This scale represents the total achieved appointments and total scheduled appointments. Data was collected weekly and added up per month.The minimum is 0 ( no appointments ) with no maximum (participants were not limited to the number of appointments per week).
Time Frame: Every week for up to 52 weeks
Measure: Mean (Standard Deviation); unit: appointments
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 55 | 55
appointments
  Total Scheduled Month 1 | 6.33 (4.25) | 3.42 (4.31)
  Total Scheduled Month 2 | 8.64 (5.59) | 4.65 (5.62)
  Total Scheduled Month 3 | 8.09 (6.26) | 4.67 (5.32)
  Total Scheduled Month4 | 7.65 (5.69) | 5.6 (6.12)
  Total Scheduled Month 5 | 6.31 (6.36) | 4.33 (5.56)
  Total scheduled Month 6 | 8.04 (7.35) | 5.11 (6.88)
  Total Scheduled Month 7 | 7.8 (7.40) | 5.85 (7.31)
  Total Scheduled Month 8 | 8.58 (7.07) | 5.8 (7.79)
  Total Scheduled Month 9 | 7.72 (7.04) | 4.69 (7.41)
  Total Scheduled Month 10 | 8.27 (7.36) | 5.15 (7.14)
  Total Scheduled Month11 | 7.05 (7.49) | 5.22 (7.01)
  Total Scheduled Month 12 | 6.95 (7.36) | 5.6 (7.44)
  Total Scheduled Month 13 | 7.53 (7.22) | 5.42 (8.09)
  Total Achieved Month 1 | 4.55 (3.07) | 2.14 (3.02)
  Total Achieved Month 2 | 4.33 (3.42) | 2.29 (2.74)
  Total Achieved Month 3 | 4.05 (4.21) | 2 (2.39)
  Total Achieved Month 4 | 3.93 (2.69) | 2.31 (2.73)
  Total Achieved Month 5 | 4.13 (4.32) | 2.38 (3.16)
  Total Achieved Month 6 | 5.16 (5.38) | 2.95 (4.66)
  Total Achieved Month 7 | 4.67 (5.39) | 3 (4.82)
  Total Achieved Month 8 | 5.07 (5.36) | 3.09 (5.47)
  Total Achieved Month 9 | 4.8 (5.09) | 2.91 (5.64)
  Total Achieved Month 10 | 4.53 (4.70) | 2.84 (5.54)
  Total Achieved Month 11 | 3.81 (4.56) | 2.84 (4.68)
  Total Achieved Month 12 | 3.55 (4.22) | 3.13 (5.55)
  Total Achieved Month 13 | 4.09 (4.47) | 2.91 (6.05)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; Between group comparison of total scheduled appointments from 1-13 months; Test type: Superiority; p = .04, ANCOVA; Mean Difference (Final Values) = 0.66
Statistical Analysis 2: Comparison: Peer Navigator Intervention vs Controlled; Between group comparison of total achieved appointments from 1-13 months; Test type: Superiority; p = .008, ANCOVA; Mean Difference (Final Values) = 0.61

2. Secondary Outcome: Attitudes Toward Seeking Professional Psychological Help Scale (ATSPPH)
Description: ATSPPH is a 29 item scale that has been used in more than 150 studies. The scale ranges from 1 (disagreement) to 4 (agreement). Higher overall scores reflect more positive attitudes towards help seeking. Subscales were summed to get the total of each scale. Total scores range from 29-116.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 55 | 55
units on a scale
  Baseline | 90.18 (13.42) | 91.15 (12.31)
  4 Month | 89.77 (10.36) | 89.7682 (11.65)
  8 Month | 89.62 (10.80) | 88.74 (11.67)
  12 Month | 91.04 (10.39) | 87.85 (13.07)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .135, ANCOVA; Mean Difference (Final Values) = 0.99

3. Secondary Outcome: Empowerment Scale (EMP)
Description: This widely used scale examines multiple dimensions of perceived personal empowerment in people with serious mental illness. The scale ranges from 1 (strongly agree) to 4 (strongly disagree). The lower the score, the higher level of empowerment. The total scores range from a minimum value of 4 to a maximum value of 16.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 55 | 55
units on a scale
  Baseline | 11.66 (1.29) | 11.12 (1.22)
  4 Month | 11.12 (1.53) | 10.79 (1.39)
  8 Month | 10.82 (1.31) | 10.96 (1.39)
  12 Month | 10.91 (1.19) | 10.99 (1.40)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .077, ANCOVA; Mean Difference (Final Values) = 0.99

4. Secondary Outcome: Recovery Assessment Scale (RAS)
Description: The RAS assesses five factors related to recovery from mental illness including hope and goals. The scale ranges from 1 (strongly disagree) to 5 (strongly agree). A higher score reflects greater attitudes towards recovery. The total score range is 22-110.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 55 | 55
units on a scale
  Baseline | 78.87 (10.62) | 85.33 (10.85)
  4 Month | 85.97 (10.23) | 85.79 (10.47)
  8 Month | 87.37 (9.91) | 85.52 (10.54)
  12 Month | 88.27 (9.80) | 85.28 (11.47)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .0005, ANCOVA; Mean Difference (Final Values) = 1.00

5. Secondary Outcome: Medical Outcome Study (SF-36)
Description: This a 36 item short form that is widely adopted measure of medical health outcomes in mental health services research. Each item is scored on a 0 to 100 range. Items in same scale are averaged together to create the 8 scale scores. Higher scores indicate better health. In the current study, the total score it the sum of all scales scores. The total score can range from 0 to 800.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 54 | 55
units on a scale
  Baseline | 319.84 (149.41) | 379.97 (165.37)
  4 Month | 420.23 (143.29) | 432.43 (171.31)
  8 Month | 427.52 (140.36) | 422.91 (176.97)
  12 Month | 444.91 (163.58) | 454.81 (168.48)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .060, ANCOVA; Mean Difference (Final Values) = 1.05

6. Secondary Outcome: Quality of Life Scale (QLS)
Description: The QLS is highly used in services research and comprises 6 items of various domains of independent living. The scale ranges from 1 (terrible) to 7 (delighted). The lower the score the less quality of life. The total scores range 6-42.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 55 | 55
units on a scale
  Baseline | 23.5 (6.92) | 26.01 (6.23)
  4 Month | 25.93 (5.19) | 27.12 (6.47)
  8 Month | 26.35 (5.56) | 26.39 (7.46)
  12 Month | 27.39 (5.81) | 26.37 (7.12)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .073, ANCOVA; Mean Difference (Final Values) = 1.03

7. Secondary Outcome: Availability Health Service Scale (AHSS)
Description: The scale measures the availability of health services. The scale ranges from 1 (Not at all) to 9 (Very much). The lower the score the less availability of a service. Items were summed to get the total of each scale. Score totals range from 26-234.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 49 | 53
units on a scale
  Baseline | 159.85 (42.41) | 157.46 (50.27369)
  4 Month | 185.72 (44.02) | 166.24 (49.62)
  8 Month | 189.18 (39.52) | 171.34 (46.29)
  12 Month | 195.23 (33.64) | 183.85 (45.17)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .34, ANCOVA; Mean Difference (Final Values) = 0.93

8. Secondary Outcome: Texas Christian University Health Form- Physical Health Subscale
Description: Assesses physical health in the last 4 months and Emotional/Mental Health in the last 30 days.The scale ranges from 1 (None of the time) to 5 (All of the time). The higher the score, the more health problems. Score totals on the physical health scale range 14-70.
Time Frame: Baseline (0), 4, 8, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Navigator Intervention | Controlled
Number analyzed (Participants) | 55 | 55
units on a scale
  Baseline | 48.40 (11.37) | 43.15 (11.92)
  4 Month | 41.67 (10.94) | 40.47 (10.58)
  8 Month | 42.62 (11.96) | 41.31 (11.74)
  12 Month | 40.59 (11.47) | 40.49 (12.85)
Statistical Analysis 1: Comparison: Peer Navigator Intervention vs Controlled; This statistical analysis applies from baseline to 12 month; Test type: Superiority; p = .21, ANCOVA; Mean Difference (Final Values) = 0.95

ADVERSE EVENTS:
Arm/Group | Peer Navigator Intervention | Controlled
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

LIMITATIONS AND CAVEATS:
Concerns to US Immigration and Customs Enforcement for those with undocumented residency status make some Latinos suspicious of institutions.Heterogeneity may influence solutions to health care concerns of these Latinos with serious mental illness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No